CLINICAL TRIAL: NCT01157702
Title: An Open-Label Phase 3 Study to Assess the Immunogenicity and Safety of a Vero Cell-Derived Trivalent Seasonal Influenza Vaccine, Strain Composition 2010/2011, in an Adult and Elderly Population
Brief Title: Yearly Strain Variation Study, 2010/2011
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 721001; 2010-020026-17 (EudraCT Number)
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Influenza; Seasonal Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Experimental): Vaccination with one dose (0.5 mL) of inactivated influenza vaccine
  Interventions: Biological: Inactivated influenza vaccine (split virus, Vero cell-derived)

INTERVENTIONS:
Biological: Inactivated influenza vaccine (split virus, Vero cell-derived) — One 0.5 mL dose of inactivated influenza vaccine in a pre-filled syringe, administered by intramuscular injection into the musculus deltoideus in the upper arm
  Other Names: Preflucel

SUMMARY:
The purpose of the study is to verify the immunogenicity and tolerance of a trivalent seasonal influenza vaccine with strain composition according to WHO/EU recommendation for the 2010/2011 season for yearly licensing application.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 59 years of age, inclusive, at the time of screening (for Stratum A only)
* Subject is 60 years of age or older, inclusive, at the time of screening (for Stratum B only)
* Subject has given written informed consent prior to study entry
* Subject is generally healthy, as determined by the investigator's clinical judgment through collection of medical history and performance of a physical examination, such that the investigator would not hesitate to provide routine influenza immunization to the subject in the course of routine medical practice
* Subject agrees to keep a daily record of symptoms for the duration of the study
* If subject is of childbearing potential, subject presents with a negative urine pregnancy test, and agrees to employ adequate birth control measures for the duration of the study
* Subject is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Subject has a history of severe allergic reaction or anaphylaxis
* Subject has an oral temperature of >= 37.5°C on the day of vaccination in this study.
* Subject has a rash or dermatologic condition or tattoos, which may interfere with injection site reaction rating
* Subject has received a live vaccine within 4 weeks or an inactivated or subunit vaccine within 2 weeks of study entry
* Subject has received a seasonal influenza vaccine within 6 months of study entry
* Subject currently has or had a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder
* Subject has any inherited or acquired immunodeficiency
* Subject has a disease or is currently undergoing a form of treatment or was undergoing a form of treatment within 30 days prior to study entry that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (>800 µg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs.
* Subject has a functional or surgical asplenia
* Subject has a known or suspected problem with alcohol or drug abuse
* Subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study.
* Subject is pregnant or lactating at the time of enrollment
* Subject has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To assess the immunogenicity to each of the three antigens contained in a trivalent seasonal influenza vaccine with strain composition according to WHO/EU recommendation for the 2010/2011 season in an adult and elderly population | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic for Clinical Pharmacology, General Hospital Vienna, Vienna, Austria